CLINICAL TRIAL: NCT00444652
Title: Thromboprophylaxis During Bariatric Surgery
Brief Title: Thromboprophylaxis and Bariatric Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: French State (Unknown); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3779
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Thromboembolism
Keywords: Thromboprophylaxis; Bariatric surgery; prevention of venous thromboembolism in bariatric surgery
MeSH Terms: conditions — Thromboembolism | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Enoxaparin — injection of enoxaparin a few time

SUMMARY:
This trial is an assessment of the efficacy of three thromboprophylaxis regimens in two types of bariatric surgery.

- gastric banding and gastric bypass on anti-Xa activity levels

The study includes two groups of 150 patients scheduled for gastric banding or gastric bypass.

Assessment of anti-Xa levels before and 4 hours after the injections from day 0 to 2 in order to determine the best prophylactic regimen allowing expected values ranged between 0.3 and 0.5 IU / ml.

ELIGIBILITY:
Inclusion Criteria:

* BMI over 40
* Gastric banding or gastric bypass

Exclusion Criteria:

* Renal insufficiency
* Thrombopenia
* Long term anticoagulant treatment
* Pregnancy
* Allergy to heparin

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-11; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Anti-Xa activity level measured 4 hours before and after enoxaparin injection at different doses | 48 heures

SECONDARY OUTCOMES:
Microparticles | day 0, 1, 9,30
Thrombotic events until D30 | day 30
Bleeding events | day 30

CONTACTS AND LOCATIONS:
Overall Officials: Annick Steib, MD, Study Director — Hôpitaux Universitaire de Strasbourg
Locations (10):
- France (10):
  - Clinique de l'Orangerie, Strasbourg, Alsace
  - Département d'Anesthésiologie Hôpital Civil, Strasbourg, Alsace
  - Laboratoire d'hémostase Hôpital de Hautepierre, Strasbourg, Alsace
  - Service de Chirurgie Digestive Hopital de Hautepierre, Strasbourg, Alsace
  - Service de Chirurgie Générale et Endocrinienne Hôpital Civil, Strasbourg, Alsace
  - Département d'Anesthésiologie Hôpital de Brabois, Nancy, Lorraine
  - Laboratoire d'Hémostase Hôpital de Brabois, Nancy, Lorraine
  - Service de Chirurgie Digestive Hôpital de Brabois, Nancy, Lorraine
  - Service de chirurgie générale et digestive,Hôpital Hôtel Dieu, Nantes
  - Centre investigation Clinique Hôpital Civil, Strasbourg

REFERENCES:
- [Derived] Amaral FC, Baptista-Silva JC, Nakano LC, Flumignan RL. Pharmacological interventions for preventing venous thromboembolism in people undergoing bariatric surgery. Cochrane Database Syst Rev. 2022 Nov 22;11(11):CD013683. doi: 10.1002/14651858.CD013683.pub2. PMID 36413425